CLINICAL TRIAL: NCT06877221
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Trial to Evaluate the Effectiveness and Safety of an Ultrasound Renal Denervation Catheter in Combination With an Ultrasound Renal Denervation Device for the Treatment of Refractory Hypertension or Drug - Intolerant Hypertension
Brief Title: Safety and Efficacy of Modulated Ultrasound Renal Denervation for HTN
Acronym: ModulationHTN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Pulsecare Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW-URDN202501
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Refractory Hypertension or Drug-intolerant Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound renal denervation (Experimental)
  Interventions: Procedure: ultrasound renal denervation
- Renal arteriography (Sham Comparator)
  Interventions: Procedure: ultrasound renal denervation

INTERVENTIONS:
Procedure: ultrasound renal denervation — Treat with an ultrasound nerve ablation catheter and an ultrasound nerve ablation device

SUMMARY:
Prospective, multicenter, randomized, controlled, blinded, and superiority - designed; The target population undergoes a screening treatment with prescribed medications for at least 4 weeks. Eligible subjects are randomly assigned to the experimental group and the control group at a ratio of 2:1. The experimental group is treated with the ultrasound nerve ablation catheter and the ultrasound nerve ablation device of Shenzhen Maiwei Medical Technology Co., Ltd., while the control group only undergoes renal arteriography (regarded as a sham operation). Within 6 months after the operation, both groups continue to receive antihypertensive drug treatment with the dosage and types specified during the screening period. The subjects are kept blinded during the study. The relative change values of the average 24 - hour ambulatory systolic blood pressure from the baseline at 6 months after the operation are compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old (calculated based on the date of starting standardized medication).
2. After treatment with at least two types of antihypertensive drugs for 4 weeks or more, the clinic systolic blood pressure is ≥140 mmHg and ≤180 mmHg, and the average 24 - hour ambulatory systolic blood pressure is ≥130 mmHg (or the daytime ambulatory systolic blood pressure is ≥135 mmHg).
3. Resting heart rate ≥70 beats per minute without taking beta - blockers (this criterion does not apply to patients taking beta - blockers).
4. The subject agrees to participate in this clinical trial, complies with the follow - up required by the trial protocol, and has voluntarily signed the informed consent form

Exclusion Criteria:

1. CTA, MRA, or DSA examination shows that the shape and structure of the unilateral or bilateral renal arteries are not suitable for ablation surgery (renal artery stenosis exceeding 50%, renal artery aneurysm, fibromuscular dysplasia of the renal artery, or the diameter of the main renal artery is less than 3 mm).
2. Having only one kidney or having received a kidney transplant.
3. Having a history of renal artery interventional treatment or renal denervation surgery.
4. Suffering from any condition that may affect the accuracy of blood pressure measurement, such as the upper arm diameter being too large relative to the cuff.
5. Secondary hypertension (excluding apnea syndrome).
6. Glomerular filtration rate (eGFR) < 45 mL/min/1.73m² (MDRD formula).
7. Having a history of hospitalization due to hypertensive crisis within one year before randomization for enrollment.
8. Suffering from type 1 diabetes.
9. Suffering from primary pulmonary hypertension.
10. Being allergic to contrast agents.
11. Severe cardiac valve stenosis.
12. Cardiac insufficiency (NYHA class III - IV).
13. Hyperthyroidism or hypothyroidism.
14. Requiring mechanical ventilation for assisted breathing (except for nocturnal respiratory support for treating sleep apnea).
15. Acute or severe systemic infection.
16. Having an implantable cardioverter - defibrillator (ICD) or pacemaker.
17. Having obvious symptoms of active peptic ulcer (such as abdominal pain, nausea, vomiting, regurgitation, etc.).
18. Having obvious bleeding tendency and hematological diseases.
19. Having a history of surgery or trauma requiring hospitalization within 30 days before randomization for enrollment.
20. Having a cardiovascular event (stable or unstable angina, myocardial infarction) or cerebrovascular event (stroke, cerebrovascular accident, transient ischemic attack) within 6 months before randomization for enrollment.
21. Pregnant, lactating women, or women planning to become pregnant during the study period.
22. Currently participating in other clinical trials of drugs or medical devices.
23. Other reasons that the investigator deems inappropriate for participation in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The average change value of 24 - hour ambulatory systolic blood pressure (ASBP) relative to the baseline | Six months after surgery
  The average change value of 24 - hour ambulatory systolic blood pressure (ASBP) relative to the baseline at 6 months after surgery

SECONDARY OUTCOMES:
The change values of clinic systolic blood pressure and diastolic blood pressure relative to the baseline | 3 months and 6 months after surgery
  The changes in clinic systolic and diastolic blood pressures relative to the baseline at 3 months and 6 months after surgery
The attainment rate of clinic diastolic blood pressure | 3 months and 6 months after surgery
  The attainment rate of clinic systolic blood pressure (90 mmHg ≤ SBP < 140 mmHg) at 3 months and 6 months after surgery The attainment rate of clinic systolic blood pressure (90 mmHg ≤ SBP < 140 mmHg) at 3 months and 6 months after surgery The attainment rate of clinic systolic blood pressure (90 mmHg ≤ SBP < 140 mmHg) at 3 months and 6 months after surgery
The average change value of 24 - hour ambulatory diastolic blood pressure relative to the baseline | 3 months and 6 months after surgery
  The average change values of 24 - hour ambulatory diastolic blood pressure relative to the baseline at 3 months and 6 months after surgery
The average change value of 24 - hour ambulatory systolic blood pressure relative to the baseline | Three months after surgery
  The average change value of 24 - hour ambulatory systolic blood pressure relative to the baseline at 3 months after surgery
The proportion of patients with a reduction in clinic systolic blood pressure of ≥5 mmHg, 10 mmHg, 15 mmHg, and 20 mmHg | 3 months and 6 months after surgery
  The proportion of patients with a reduction in clinic systolic blood pressure of ≥ 5 mmHg, 10 mmHg, 15 mmHg, and 20 mmHg at 3 months and 6 months after surgery
Changes in the drug composite index of the types and dosages of antihypertensive medications | Six months after surgery
  Changes in the drug composite index of the types and dosages of antihypertensive drugs 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No